CLINICAL TRIAL: NCT00551525
Title: A Phase II Trial of Samarium 153 Followed by Salvage Prostatic Fossa 3D-CRT or IMRT Irradiation in High-Risk, Clinically Non-Metastatic Prostate Cancer After Radical Prostatectomy
Brief Title: Samarium Sm 153 Lexidronam Pentasodium and 3-Dimensional Conformal Radiation Therapy or Intensity-Modulated Radiation Therapy in Treating Patients With Rising Prostate-Specific Antigen Levels After Radical Prostatectomy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0622; CDR0000570622; NCI-2009-01094 (Registry Identifier: CTRP(Clinical Trial Reporting Program)); NCT01317043 (obsolete NCT alias)
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Samarium-153; samarium Sm-153 lexidronam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy + Samarium 153 (Experimental): Samarium 153 infusion followed by radiotherapy 12 weeks later
  Interventions: Radiation: Radiotherapy; Drug: Samarium 153

INTERVENTIONS:
Radiation: Radiotherapy — 3D-CRT or IMRT 64.8-70.2 Gy to the prostatic fossa begins 12 weeks (+/- 1 week) after Samarium 153 administration. Daily tumor doses of 1.8 - 2.0 Gy per day, 5 days per week x 7-8 weeks.
  Other Names: 3D-CRT; IMRT; Intensity-modulated radiation therapy
Drug: Samarium 153 — Samarium 153 lexidronam dose 2.0 mCi/kg by IV injection one time within 2 weeks (+/- 3days) after registration.
  Other Names: Samarium sm 153 lexidronam pentasodium; Quadramet

SUMMARY:
RATIONALE: Giving samarium Sm 153 lexidronam pentasodium and 3-dimensional (3-D) conformal radiation therapy or intensity-modulated radiation therapy may keep prostate cancer from growing in patients with rising prostate-specific antigen (PSA) levels after radical prostatectomy for prostate cancer.

PURPOSE: This phase II trial is studying how well samarium Sm 153 lexidronam pentasodium and 3-D conformal radiation therapy or intensity-modulated radiation therapy work in treating patients with rising PSA levels after radical prostatectomy for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the effectiveness of samarium Sm 153 lexidronam pentasodium (as determined by a 30% decline in the PSA level within 12 weeks) followed by either three-dimensional conformal radiation therapy or intensity-modulated radiation therapy in patients with rising prostate-specific antigen levels (PSA) after radical prostatectomy prostate cancer.

Secondary

* To assess the proportion of patients completing protocol treatment.
* To evaluate hematological toxicity at 12 weeks.
* To evaluate samarium Sm 153 lexidronam pentasodium-related adverse events at 12 weeks.
* To evaluate the "acute" and "late" radiation therapy-related events having occurred up to 24 weeks from the end of radiation therapy.
* To compare the freedom from progression rate at 2 years to that predicted by the Kattan Nomograms.

OUTLINE: Patients receive samarium Sm 153 lexidronam pentasodium (SM) IV on day 1. Patients are closely monitored for prostate-specific antigen (PSA) level and SM-associated toxicity for 12 weeks. After the 12 weeks, patients undergo either intensity-modulated radiation therapy or 3-dimensional conformal radiation therapy 5 days a week for 7-8 weeks. Patients may receive hormonal therapy (after radiation therapy) at the discretion of their physician.

Treatment continues in the absence of disease progression (defined as a PSA doubling time less than 3 months), severe thrombocytopenia (defined as a platelet count of 25,000 cells/mm³ or less), or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3 months, 6 months, and 12 months, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically proven diagnosis of prostate cancer progressing after prior radical prostatectomy as indicated by one of the following:

  * Postoperative prostate-specific antigen (PSA) rising above 1.0 ng/mL
  * Postoperative PSA rising above 0.2 ng/mL with a surgical tumor Gleason score of 9 or 10
  * Postoperative PSA rising above 0.2 ng/ml with nodal disease
* Stage II-IV disease (T2 -T4, N0-N1)
* No distant metastases based on the following minimum diagnostic work up:

  * History or physical examination within the past 8 weeks
  * Bone scan negative for bone metastases within the past 4 months
  * Abdominal imaging negative for metastases within the past 6 months

Exclusion criteria:

* Biopsy evidence of M1 disease
* Presence of neuroendocrine features in any prostate cancer specimen

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Zubrod Performance Status 0-1
* Absolute neutrophil count (ANC) ≥ 1,800 cells/mm³
* Platelet count ≥ 100,000 cells/mm³
* Hemoglobin ≥ 8.0 g/dL (transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is permitted)

Exclusion criteria:

* Prior invasive malignancy (except nonmelanoma skin cancer) unless disease free for a minimum of 3 years
* Severe, active comorbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects (laboratory tests for liver function and coagulation parameters, however, are not required for entry into this protocol)
  * Renal failure (laboratory tests for renal function, however, are not required for entry into this protocol)
  * AIDS based upon current Centers for Disease Control (CDC) definition (HIV testing is not required)

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy for the study cancer

  * Prior chemotherapy for a different cancer is permitted
* No hormonal therapy initiated within the last 3 months
* No prior radiotherapy to the pelvic region that would result in overlap of radiotherapy fields

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-04; Primary Completion 2014-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K. Valicenti, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University; Oliver Sartor, MD, Study Chair — Dana-Farber Cancer Institute
Locations (29):
- United States (29):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Solano Radiation Oncology Center, Vacaville, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - Stony Brook University Cancer Center, Stony Brook, New York
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Robinson Radiation Oncology, Ravenna, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Coastal Cancer Center at Sentara Virginia Beach General Hospital, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiotherapy + Samarium 153
Started | 67
Completed | 62 (Subjects with data available for analysis are considered to have completed the study)
Not Completed | 5
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Population: All eligible patients
Arm/Group | Radiotherapy + Samarium 153
Number analyzed (Participants) | 62
Age, Continuous [Median (Full Range); unit: years] | 65 [49 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 62

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With PSA Response (pt) Within 12 Weeks of Samarium 153 Administration
Description: A PSA response for each patient is calculated by (baseline PSA-current PSA)/baseline PSA. A decline of at least 30% is considered a response. Null hypothesis (H0): Samarium 153 is not effective (pt ≤ 0.1) vs alternative hypothesis (HA): Samarium 153 is effective (pt ≥ 0.25). The sample size of 69 analyzable patients (eligible patients receiving any protocol treatment with ≥ 12 weeks follow-up from the Samarium 153 injection) was calculated based on Fleming's Multiple Testing Procedure at a significance level of 0.019 and 91% statistical power requiring 69 patients to conclude either the null or alternative hypotheses. With only 52 analyzable patients this study had only 78% power and needed at least 11 patients with a PSA response to reject H0.
Time Frame: Twelve weeks from the date of Samarium 153 infusion.
Population: All eligible patients who received Samarium 153 with at least 12 weeks follow-up from the injection
Measure: Number; unit: percentage of participants
Arm/Group | Radiotherapy + Samarium 153
Number analyzed (Participants) | 52
percentage of participants | 7

2. Secondary Outcome: Completion of Therapy
Description: The completion of protocol treatment is defined as receiving at least 64.8 Gy radiation after the Samarium 153 injection. The null hypothesis that the proportion of the number of patients who complete the protocol treatment (the Samarium 153 and the radiation therapy) is less than or equal to 0.5 was tested using an exact test for a binomial proportion. If the true treatment completion proportion is 0.8, then the statistical power of a one-sided 0.378 level exact binomial test of proportion would be 94.1% with the sample size of 26. Therefore any number of analyzable patients greater than 26 patients provides enough power for this endpoint.
Time Frame: 90 days from the end of radiation therapy.
Population: All eligible patients who started treatment and did not withdraw consent prior to 90 days from the end of radiation therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy + Samarium 153
Number analyzed (Participants) | 60
percentage of participants | 93.3 [87.0 to 99.7]
Statistical Analysis 1: Comparison: Radiotherapy + Samarium 153; Test type: Superiority or Other; p < 0.001, binomial proportion — Significance level 0.05, two-sided test

3. Secondary Outcome: Number of Patients With Hematologic Toxicity at 12 Weeks
Description: Adverse events are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. Hematological toxicities consist of platelet grade 3-5, white blood cell grade 3-5, hemoglobin grade 3-5, and any secondary leukemia's.
Time Frame: Twelve weeks from the date of Samarium 153 infusion.
Population: Eligible patients who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy + Samarium 153
Number analyzed (Participants) | 60
Participants | 15

4. Secondary Outcome: Samarium 153-related Adverse Events at 12 Weeks (Percentage of Patients)
Description: Adverse events are evaluated by the NCI Common Terminology Criteria for Adverse Event (CTCAE) version 3.0. The treatment-related attribution includes definitely, probably or possibly related to treatment. The treatment-related adverse events are:
  * HEMATOLOGIC Platelet grade 3-5 White blood cell count (WBC) grade 3-5 Hemoglobin grade 3-5 Any secondary leukemia's
  * HEMORRHAGE/BLEEDING Hemorrhage, gastrointestinal - anus, rectum grade 3-5 Hemorrhage, genitourinary - bladder, prostate, urethra grade 3-5
  * SAMARIUM 153-RELATED GRADE 5 ADVERSE EVENT PRIOR TO TREATMENT OF RADIATION.
Time Frame: Twelve weeks from the date of Samarium 153 infusion
Population: Eligible patients with adverse event data
Measure: Number; unit: percentage of participants
Arm/Group | Radiotherapy + Samarium 153
Number analyzed (Participants) | 60
percentage of participants | 16

5. Secondary Outcome: Acute and Late Radiotherapy-Related Adverse Events
Description: The number of patients who experienced a grade 1-5 radiation-related adverse events within 90 days of the start of radiotherapy (acute) and after 90 days (late). Adverse events are evaluated by the NCI Common Terminology Criteria for Adverse Event (CTCAE) version 3.0. Multivariate logistic regression was used to model the association of clinical T-stage (pT2 vs. pT3 [reference level]), baseline PSA, Gleason score (<8 vs. 8-10[reference level]), and age with the occurrence of any acute radiotherapy-related adverse event. Odds ratios and the respective 95% confidence intervals were computed for each factor. Per the protocol, late adverse events were not analyzed.
Time Frame: 90 days from start of radiotherapy
Population: Eligible patients with adverse event data
Measure: Number; unit: participants
Arm/Group | Radiotherapy + Samarium 153
Number analyzed (Participants) | 60
participants
  Acute | 35
  Late | 27
Statistical Analysis 1: Comparison: Radiotherapy + Samarium 153; Modeling the association of age with the occurrence of any acute radiotherapy-related adverse event, adjusting for clinical T-stage (pT2 vs. pT3 [reference level]), baseline PSA, and Gleason score (<8 vs. 8-10[reference level]); Test type: Superiority or Other; Odds Ratio (OR) = 0.984, 95% CI 2-sided [0.910 to 1.063]
Statistical Analysis 2: Comparison: Radiotherapy + Samarium 153; Modeling the association of baseline PSA with the occurrence of any acute radiotherapy-related adverse event, adjusting for clinical T-stage (pT2 vs. pT3 [reference level]), Gleason score (<8 vs. 8-10[reference level]), and age; Test type: Superiority or Other; Odds Ratio (OR) = 1.020, 95% CI 2-sided [0.890 to 1.169]
Statistical Analysis 3: Comparison: Radiotherapy + Samarium 153; Modeling the association of clinical T-stage (pT2 vs. pT3 [reference level]) with the occurrence of any acute radiotherapy-related adverse event, adjusting for baseline PSA, Gleason score (<8 vs. 8-10[reference level]), and age; Test type: Superiority or Other; Odds Ratio (OR) = 1.307, 95% CI 2-sided [0.364 to 4.697]
Statistical Analysis 4: Comparison: Radiotherapy + Samarium 153; Modeling the association of Gleason score (<8 vs. 8-10[reference level]) with the occurrence of any acute radiotherapy-related adverse event, adjusting for clinical T-stage (pT2 vs. pT3 [reference level]), baseline PSA, and age; Test type: Superiority or Other; Odds Ratio (OR) = 0.659, 95% CI 2-sided [0.217 to 2.006]

6. Secondary Outcome: Freedom From Progression (FFP) Rate at 2 Years
Description: Progression is defined as biochemical (PSA) failure at any time for 2 years after prostatic fossa radiation therapy (RT), initiation of systemic therapy, or clinical failure. Biochemical failure is defined as a rise of 0.2 ng/ml or more above the nadir PSA after completion of RT followed by another higher value, or a continued rise in the serum PSA despite RT. FFP rate at 2 years was to be compared to that predicted by the Kattan Nomograms. See "Limitations and Caveats" section.
Time Frame: From randomization to 2 years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy + Samarium 153
Number analyzed (Participants) | 60
percentage of participants | 25.50 [14.40 to 36.70]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event. Eligible patients with any adverse event data are included.
Arm/Group | Radiotherapy + Samarium 153
Serious Adverse Events (participants affected / at risk) | 5/60
Other Adverse Events (participants affected / at risk) | 55/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy + Samarium 153 (N=60)
Sudden death (General disorders) | 1
Leukopenia (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy + Samarium 153 (N=60)
Blood disorder (Blood and lymphatic system disorders) | 7
Hemoglobin decreased (Blood and lymphatic system disorders) | 25
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 15
Gastrointestinal disorder (Gastrointestinal disorders) | 9
Hemorrhoids (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 6
Proctitis (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 30
Pain [other] (General disorders) | 3
Alanine aminotransferase increased (Investigations) | 3
Leukopenia (Investigations) | 39
Lymphopenia (Investigations) | 11
Neutrophil count decreased (Investigations) | 26
Platelet count decreased (Investigations) | 46
Hyperglycemia (Metabolism and nutrition disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Urinary frequency (Renal and urinary disorders) | 26
Urinary incontinence (Renal and urinary disorders) | 16
Urinary retention (Renal and urinary disorders) | 4
Urogenital disorder (Renal and urinary disorders) | 10
Erectile dysfunction (Reproductive system and breast disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 3
Hot flashes (Vascular disorders) | 10

LIMITATIONS AND CAVEATS:
Comparison of freedom from progression rate at two years with Kattan Nomograms was not possible because the pretreatment data needed for the Kattan Nomograms was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.